CLINICAL TRIAL: NCT00004938
Title: Phase II Study of Fluconazole for Lymphocutaneous and Visceral Sporotrichosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11815; NIAID-MSG-11815
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2000-04

CONDITIONS: Sporotrichosis
Keywords: fungal infection; rare disease; sporotrichosis
MeSH Terms: conditions — Sporotrichosis; Mycoses; Rare Diseases | interventions — Fluconazole

INTERVENTIONS:
Drug: fluconazole

SUMMARY:
OBJECTIVE:

I. Evaluate the efficacy of fluconazole in patients with lymphocutaneous or visceral sporotrichosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are treated with daily oral fluconazole for up to 24 months. Follow-up continues for at least 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Presumptive evidence of sporotrichosis Culture-proven sporotrichosis determined on study Relapsing disease following antifungal therapy eligible if culture positive for Sporothrix schenckii prior to entry No life-threatening disease No central nervous system sporotrichosis --Prior/Concurrent Therapy-- No concurrent drugs known to react with fluconazole No more than 3 days of systemic antifungals for current sporotrichosis episode --Patient Characteristics-- Hepatic: Liver function tests no greater than 5 times normal Other: No HIV infection No pregnant or nursing women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1996-08; Study Completion 1996-08

CONTACTS AND LOCATIONS:
Overall Officials: William Dismukes, Study Chair — University of Alabama at Birmingham

REFERENCES:
- [Background] Kauffman CA, Pappas PG, McKinsey DS, Greenfield RA, Perfect JR, Cloud GA, Thomas CJ, Dismukes WE. Treatment of lymphocutaneous and visceral sporotrichosis with fluconazole. Clin Infect Dis. 1996 Jan;22(1):46-50. doi: 10.1093/clinids/22.1.46. PMID 8824965